CLINICAL TRIAL: NCT05770947
Title: Cognitive Behavioral Therapy for Adolescents With Bulimia Nervosa and Higher Weight (Online Treatment Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Eating Disorders Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000033150
Record Dates: First submitted 2023-03-03; First posted 2023-03-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bulimia Nervosa; Overweight or Obesity
MeSH Terms: conditions — Bulimia Nervosa; Overweight; Obesity | interventions — Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy for adolescents with higher weight seeking treatment for bulimia nervosa (CBT-BNh).Designed for adolescents, CBT-BNh will include psychoeducation, cognitive restructuring, and relapse prevention planning. The focus of therapy will include reducing extreme/unhealthy weight-control behaviors (purging) as well as binge eating, and self-compassion coping skills will address weight stigma and self-directed weight criticism.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Mindfulness (Active Comparator): Learning to Breathe (L2B) is an existing, evidence-based program for adolescents that teaches mindfulness skills each week, including time to practice and reflect. the skills are grouped into six themes: Body, Reflections, Emotions, Attention, Tenderness, Habits, and Empowerment.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) is a psychological treatment or "talk therapy" that integrates how people think, feel, and behave to create new behavior patterns that improve thinking processes and reduce distress.
  Arms: Cognitive Behavioral Therapy
Behavioral: Mindfulness — Mindfulness is a psychological treatment or "talk therapy" that practices different coping skills to improve thinking processes and reduce distress.
  Other Names: Learning to Breathe
  Arms: Mindfulness

SUMMARY:
This study will test the feasibility and acceptability of two treatments for adolescents with higher weight seeking treatment for bulimia nervosa (binge eating and purging, or going to extremes to lose weight).

DETAILED DESCRIPTION:
This study will test the feasibility and acceptability of two treatments for adolescents with higher weight seeking treatment for bulimia nervosa. Bulimia nervosa is when individuals binge eat (overeat while feeling like they lost control) and purge (do something extreme or unhealthy to lose weight or prevent weight gain). Bulimia nervosa happens across different ages and body sizes. This study is focusing on adolescents who have a larger body size. Adolescents will receive treatment that is 4 months of 45-minute sessions, weekly. Treatment will occur over telehealth (e.g., zoom), and the whole study is online.

ELIGIBILITY:
Inclusion Criteria:

* Have higher weight (>85th BMI percentile or >85th percentile in past year)
* 2 binge/purge episodes per month for the prior 3 months
* Be otherwise-healthy youth (i.e., no uncontrolled or serious medical conditions);
* Read, comprehend, and write English at a sufficient level to complete study-related materials;
* Provide an approval form from a healthcare provider;
* Provide a signed and dated written assent (or consent for youth age 18 or 19) prior to study participation;
* Provide a signed and dated written consent from one parent prior to study participation;
* Be available for participation in the study for 4 months.

Exclusion Criteria:

* Medical or psychiatric conditions requiring hospitalization or intensive care
* anorexia nervosa
* developmental or cognitive disorders that would interfere with therapy
* pregnancy or breastfeeding
* concurrent treatments (medication or psychological) influencing appetite or weight
* began hormone therapy in prior 3 months

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Bulimia nervosa remission assessed by the Eating Disorder Examination Questionnaire (EDE-Q) | baseline and post-treatment (Month 4)
  Remission from binge eating and purging behaviors will be assessed by EDE-Q. The EDE-Q is a self-report questionnaire with four subscales and a global severity score. the global score ranges from 0-6 with higher scores reflecting greater severity of eating disorder behaviors.

SECONDARY OUTCOMES:
Change in Binge eating frequency assessed by the EDE-Q | baseline and post-treatment (Month 4)
  Number of episodes of binge eating in past month
Change in Purging frequency assessed by the EDE-Q | baseline and post-treatment (Month 4)
  Number of episodes of purging in past month
Change in eating disorder psychopathology assessed by the Eating Disorder Examination Questionnaire (EDE-Q) global score. | baseline and post-treatment (Month 4)
  Eating disorder psychopathology will be assessed using the EDE-Q global score. The EDE-Q is a self-report questionnaire with four subscales and a global severity score. the global score ranges from 0-6 with higher scores reflecting greater severity of eating disorder psychopathology.
Change in Depression assessed using Patient Health Questionnaire-9 (PHQ-9) | baseline and post-treatment (Month 4)
  Depression will be assessed using the PHQ-9. PHQ-9 is a validated questionnaire used to screen for depression with a range of scores from 0-27. Higher scores indicate more severe depressive symptoms.
Change in Self-esteem assessed using the Rosenberg Self-Esteem Scale (RSES) | baseline and post-treatment (Month 4)
  Self-esteem will be assessed using the RSES. The RSES is a self-report measure that consists of 10 statements related to overall feelings of self-worth or self-acceptance. The items are answered on a four-point scale ranging from strongly agree to strongly disagree. The total score ranges from 0 to 30 with higher scores indicating higher self esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Lydecker, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University (Teen Power - Online), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Because of the sensitive nature of these data, IPD sharing will be limited to requests from other researchers that are reasonable and accompanied by an approved protocol.